CLINICAL TRIAL: NCT04245683
Title: Feasibility of Non-Operative Management of Rectal Cancer in a Rural Population
Status: Recruiting | Type: Observational
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Eric Bravin, attending physician - medical oncology, Bassett Healthcare
Other Study IDs: 1526939
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative Group: Patients who select operative treatment and follow up after successful neoadjuvant treatment.
  Interventions: Procedure: Bowel/rectal resection
- Non-operative Group: Patients who select non-operative follow up after successful neoadjuvant treatment
  Interventions: Other: non-operative follow up

INTERVENTIONS:
Procedure: Bowel/rectal resection — surgical removal of the portion of the rectum where the tumor was originally identified
  Groups: Operative Group
Other: non-operative follow up — patients who choose the non-operative option will be required to adhere to a very intensive follow up protocol, including endoscopy and CT imaging
  Groups: Non-operative Group

SUMMARY:
This is an observational research study. Patients with rectal cancer can choose different courses of treatment. This study will follow these patients over the course of approximately six years, depending on their treatment. Patients will be monitored through clinic visits and survey assessments to see how they do, how they feel regarding their treatment choices, and their outcomes. The surveys will analyze the impact of the patients' treatment choices, as well as patient adherence, in a rural setting.

DETAILED DESCRIPTION:
Standards of care for patients with rectal cancer are evolving over time. Surgery for rectal cancer is associated with significant short- and long-term side effects for patients, including changes in bowel function, self-image, ability to work, and sexual function. Emerging data indicates that some patients experiencing complete clinical response to neoadjuvant therapy (treatment given prior to surgery) may be able to forego surgery, without compromising cancer outcomes. Current National Cancer Center Network (NCCN) guidelines for the treatment of rectal cancer states that, "...the panel believes that a non-operative management approach may be considered in centers with experienced multi-disciplinary teams, after a careful discussion with the patient of his or her risk tolerance." Between 15-27% of patients achieve a complete pathological response after chemoradiotherapy (CRT), which is administered before surgery, and have low rates of local recurrence and high rates of overall survival. Treating these patients without surgery has been a focus in recent years. Supporting data is mainly from large academic institutions, which have pioneered the approach. There is very little data on this approach in rural populations. While this approach is not considered to represent the standard of care, increasing numbers of patients are choosing to pursue it. It would be useful to accumulate data on treatment of rectal cancer in a rural setting.

The study will collect and analyze data on patient preference for operative versus non-operative management, as well as patient adherence to the careful surveillance regimen required for those electing nonoperative management. In addition, patient outcomes with a focus on quality of life, as measured on a standardized tool at multiple points before, during, and after treatment will be analyzed.

Patients will undergo an initial staging evaluation, regardless of study consent, to include:

* Physical examination
* Endoscopy
* CEA, CBC, CMP
* Pelvic MRI +/- IV contrast preferred, or if MRI contraindicated, endoscopic ultrasound
* CT Chest/Abdomen/Pelvis

Patients will also complete the following survey assessments at the time of study consent:

* Pain Assessment
* QOL- CR29
* QOL- C30
* QOL- Patient Satisfaction Survey

Patients with potentially resectable, newly diagnosed, rectal cancer will receive one of three treatment protocols based on patient and physician preference. These treatment options are considered normal standard of care and are available to all patients regardless of study participation.

Treatment choices are:

1. 5-Fluorouracil or Capecitabine with radiotherapy for 6 weeks, followed by a break of 8-12 weeks. Patients who elect this treatment plan will be reevaluated/restaged as described below, then will receive an additional 18 weeks of chemotherapy. Depending on the patient's decision regarding surgery, chemotherapy will be initiated either 4 weeks post-operatively or immediately after restaging for patients electing to forgo surgery.
2. Total Neoadjuvant Therapy (TNT) option 1: 6 cycles of Leucovorin Calcium, Fluorouracil, and Oxaliplatin (FOLFOX) over 12 weeks, followed by 6 weeks 5-Fluorouracil or Capecitabine with radiation, then a break of 10-12 weeks 3. TNT option 2: 6 weeks 5-Fluorouracil or Capecitabine with radiation, followed by 6 cycles of FOLFOX over 12 weeks, then a break of 10-12 weeks.

Patients will be monitored throughout their treatments. Treatment will be held at the discretion of the medical oncologist or radiation oncologist for severe skin reactions, severe diarrhea, severe urinary difficulty, admission to the hospital, and neutropenia with or without fever. At the completion of neoadjuvant therapy, there will be a 10-12 week observation period to allow for healing and resolution of inflammation. Patients who do not complete neoadjuvant therapy will be removed from the study. Patients who do complete neoadjuvant therapy will then undergo evaluation of their response using the modalities listed below: Physical Examination Endoscopy CEA Pelvic MRI +/- IV contrast or EUS Biopsy at surgeons discretion of residual mucosal abnormalities

Patients who do not achieve a complete tumor response would not be eligible for non-surgical management, but would continue to be followed for survival.

Those achieving complete tumor responses, as defined by no evidence of tumor on physical examination, endoscopy, MRI, and with a normal CEA value, will then have further discussion with their treating physicians regarding operative vs. non-operative management. The choice of operative or non-operative management will be left to the discretion of the physicians and the patient. Patients will also be presented at the Multidisciplinary Tumor Board to receive input on care.

After patients have been restaged, but prior to any further treatment, the following survey assessments will occur:

* Pain Assessment
* QOL- CR29
* QOL- C30
* QOL- Patient Satisfaction Survey

Operative patients will undergo surgery. They will then either complete their chemotherapy treatment if the patient has not already done so, or go directly to surveillance. Patients will be followed by surveillance for a total of 5 years post operatively. Patients will have CT imaging of the chest/abdomen/pelvis every 6-12 months for 5 years following resection, per NCCN guidelines for patients with stage II or stage III rectal cancer.

Per NCCN guidelines, non-operative patients will either complete their chemotherapy treatment if the patient has not already done so, or go directly to surveillance. Surveillance will consist of having CEA, endoscopy, and imaging (CT scans and MRI) every 3 months for 1 year; then CEA and endoscopy every 3 months with imaging (CT scans and MRI) every 6 months for the next 2 years; and then CEA and endoscopy every 6 months with imaging (CT scans and MRI) every year for 2 years.

ELIGIBILITY:
Inclusion Criteria:

For a patient to be considered eligible for this study, ALL of the following conditions must be met:

1. Age 18 or greater
2. ECOG PS 0-2
3. Stage II or III, newly diagnosed, biopsy proven, rectal cancer
4. No prior treatment for rectal cancer
5. No prior pelvic radiotherapy
6. Willing to undergo study related testing and monitoring after treatment
7. Women of childbearing potential must rule out pregnancy within 2 weeks prior to registration with a blood test or urine study
8. Women must not be pregnant or breastfeeding
9. Able to provide informed consent

Exclusion Criteria:

Patients are NOT considered eligible for this study if any of the following conditions apply:

1. Patients with metastatic disease
2. Patients that are not candidates for surgery
3. Patients that refuse neoadjuvant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with biopsy proven , resectable rectal cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
patient preferences for operative vs. non-operative management of rectal cancer | 8 months
  Number of eligible patients who select operative versus non-operative management after successfully completing approximately 20 weeks of neoadjuvant treatment and the 10-12 week post treatment observation period

SECONDARY OUTCOMES:
Patient adherence to surveillance protocols | 5 years
  Percentage of patients who choose non-operative management who successfully comply with the post-neoadjuvant treatment surveillance protocol

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bravin, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No